CLINICAL TRIAL: NCT05251181
Title: A Multi-Centric, Randomized, Double-Blind, Placebo-controlled, Phase-III Study to Assess Safety and Efficacy of Centhaquine as a Resuscitative Agent to be Used as an Adjuvant to Standard Treatment of Hypovolemic Shock
Brief Title: A Study to Assess Safety and Efficacy of Centhaquine as a Resuscitative Agent
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmazz, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Centhaquine/CT-3.2/2021
Record Dates: First submitted 2022-02-11; First posted 2022-02-22 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Hypovolemic Shock
MeSH Terms: conditions — Shock | interventions — Saline Solution; centhaquine

STUDY DESIGN:
Intervention Model Description: This is a multi-centric, randomized, double-blind, placebo-controlled phase-III clinical study to assess the safety and efficacy of centhaquine therapy in patients with hypovolemic shock with systolic arterial blood pressure ≤ 90 mmHg at presentation and continue to receive standard treatment of shock.
  This protocol is designed to develop a novel first-in-class treatment for use in critical care and life-threatening condition of hypovolemic shock with unmet need and is of national interest.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In this double-blind study, the subject and all relevant personnel involved with the conduct and interpretation of the study (including investigator, investigational site personnel, and the sponsor or designee's staff) will remain blinded to the identity of the Investigational Product (IP) assigned and the randomization codes. The final randomization list will be kept strictly confidential, filed securely by the independent biostatistician, and accessible only to authorized persons as per the sponsor's standard operating procedures until the completion of the study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Normal saline (Active Comparator): Hypovolemic shock patients will be provided the standard of care. Following randomization 100 ml (equal volume to experimental arm) of normal saline will be administered intravenously over 1 hour.
  Interventions: Drug: Normal Saline
- Centhaquine (Experimental): Hypovolemic shock patients will be provided the standard of care. Following randomization centhaquine (0.01 mg/kg) will be administered intravenously over 1 hour in 100 mL of normal saline.
  Interventions: Drug: Centhaquine

INTERVENTIONS:
Drug: Normal Saline — Normal Saline to be Used as Vehicle in the Phase-III Study to Assess Efficacy of Centhaquine as a Resuscitative Agent for Hypovolemic Shock
  Other Names: Vehicle
  Arms: Normal saline
Drug: Centhaquine — Phase-III Study to Assess Efficacy of Centhaquine as a Resuscitative Agent for Hypovolemic Shock
  Other Names: PMZ-2010
  Arms: Centhaquine

SUMMARY:
This protocol is designed to develop a novel first-in-class treatment for use in critical care and life-threatening condition of hypovolemic shock with unmet need and is of national interest. Shock is a life-threatening condition of circulatory failure. It is a state of cellular and tissue hypoxia due to reduced oxygen delivery and/or increased oxygen consumption or inadequate oxygen utilization. Shock most commonly occurs when there is circulatory failure leading to reduced tissue perfusion. There are four types of shock: distributive, cardiogenic, hypovolemic, and obstructive. However, these are not exclusive, and many patients with circulatory failure have a combination of more than one form of shock (multifactorial shock).

DETAILED DESCRIPTION:
Despite advances in medical science, treatments for hypovolemic shock have changed little in the past 30-40 years. A wounded soldier bleeding on the battlefield, or a trauma victim, is treated today largely as the patient would have been treated in 1970. The primary goal when treating traumatic hemorrhage is to control blood loss, support ventilation and oxygenation, and maintain cardiovascular function to preserve organ blood perfusion. Rapid volume repletion is indicated in patients with severe hypovolemic shock. Delayed therapy can lead to ischemic injury and possibly to irreversible shock and multiorgan system failure. Although resuscitation with intravenous fluids and blood products has remained the gold standard over the last twenty years, vigorous volume resuscitation may not be curative and has been associated with the development of serious complications including coagulopathy, acute lung injury, and abdominal compartment syndrome. Massive resuscitation also profoundly alters the neuroendocrine milieu needed to maintain vasomotor tone and may lead to a state of recalcitrant hypotension, multi-organ failure, and ultimately death in severely injured patients. Vasopressors are generally used to increase blood pressure and cardiac output, but sometimes they are not recommended since they do not correct the primary problem and tend to reduce tissue perfusion further.

This study seeks to address the impact of centhaquine on the patient population with hypovolemic shock (prehospital SBP ≤ 90 mmHg). The inclusion of centhaquine during resuscitation could potentially prevent the profound hypotension seen in late-stage shock, limit the need for aggressive volume and blood product resuscitation, and decrease the incidence of resuscitation-associated complications. This study will investigate if early use of centhaquine during the resuscitation of hypovolemic shock results in improved survival at Day 28, fewer blood transfusions, a decreased need for crystalloid resuscitation, and a lower incidence of resuscitation related complications.

In animal models of hypovolemic shock, low doses (0.006 to 0.05 mg/kg) of centhaquine proved to be highly effective in resuscitation. Centhaquine significantly decreased blood lactate and increased mean arterial pressure (MAP), pulse pressure, and cardiac output (CO), as well as decreased mortality and increased the survival time of animals with severe blood loss. Furthermore, its resuscitative effect was significantly greater compared to presently used resuscitative solutions. The proposed mechanism of action of centhaquine is that in low doses, it acts on α2B adrenergic receptors to produce venous constriction and a consequent increase in venous return to the heart, and stimulation of sodium sense in the brain to increase the intravascular blood volume. These effects increase cardiac output and tissue blood perfusion, which may be responsible for its resuscitative action.

Centhaquine has been found to be an effective resuscitative agent in rat, rabbit, and swine models of hemorrhagic shock. Its safety and tolerability have been demonstrated in a human phase I study in 25 subjects. Clinical phase II and III results indicate that centhaquine is a novel first-in-class, highly effective resuscitative agent for hypovolemic shock due to blood loss. Safety and highly significant efficacy in improving blood pressure, lactate levels, base deficit, and reduction in the use of vasopressors and reduced mortality obtained in phase II and III studies in patients of hypovolemic shock are convincing. Therefore, a phase III clinical study in the United States and Europe will be conducted in patients of hypovolemic shock patients.

The present multi-centric, randomized, double-blind, placebo-controlled phase-III study aims to assess the efficacy and safety of centhaquine as a resuscitative agent to be used as an adjuvant to standard treatment of hypovolemic shock.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in the study if he/she fulfils the following criteria:

1. Adult males or females aged 18 years or older.
2. Subjects with hypovolemic shock admitted to the hospital with systolic blood pressure ≤ 90 mm Hg at presentation, Mean Arterial Pressor (MAP) ≤ 65 mm Hg and continue to receive standard treatment of shock (endotracheal intubation; fluid resuscitation and vasopressors). Standard of care to be provided to the subject shall be the one used in that hospital.
3. Blood lactate level indicative of hypovolemic shock with lactate level more than 2 mmol/L.

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if he/she meets any of the following exclusion criteria:

1. Subject with illness clinically defined as septic shock (Procalcitonin plasma levels of ≥0.5 ng/mL) or cardiogenic shock or neurogenic shock.
2. Subject for whom an etiology for hypovolemic shock cannot be determined on initial evaluation.
3. Hypovolemic shock due to traumatic brain injury, traumatic tamponade, traumatic tension pneumothorax, ventricular wall rupture.
4. Patient with altered consciousness not due to hypovolemic shock.
5. Subject with confirmed pregnancy.
6. Cardiopulmonary resuscitation (CPR) before randomization.
7. Presence of a do not resuscitate order.
8. Patient is participating in another interventional study.
9. Patients with systemic diseases which were already present before having trauma, such as: cancer, chronic renal failure, liver failure, decompensated heart failure or AIDS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with all-cause mortality [Time frame: Day 0 through day 28]. | Day 0 through day 28
  Incidence of mortality

SECONDARY OUTCOMES:
Proportion of subjects with all-cause mortality within 48 hours | 48 hours
  Proportion of subjects with all-cause mortality within 48 hours
Change in Mean Arterial Pressure (MAP) from baseline of at least 10 mm Hg; Mean through 48 hours and at the time of discharge or day 7 | First 48 hours and at the time of discharge or day 7
  Change in Mean Arterial Pressure (MAP) from baseline of at least 10 mm Hg; Mean through 48 hours and at the time of discharge or day 7
Time (hours) to decrease blood lactate level to <2 mmol/L | 48 hours
  Time (hours) to decrease blood lactate level to <2 mmol/L; Mean through 2 hours for the first 12 hours, then every 6 hours for the next 36 hours.
Proportion of patients with adverse events (AEs) and serious adverse events (SAEs) | Day 0 through day 28
  Proportion of patients with adverse events (AEs) and serious adverse events (SAEs)

REFERENCES:
- [Background] Geevarghese M 3rd, Patel K, Gulati A, Ranjan AK. Role of adrenergic receptors in shock. Front Physiol. 2023 Jan 16;14:1094591. doi: 10.3389/fphys.2023.1094591. eCollection 2023. PMID 36726848
- [Background] Ranjan AK, Gulati A. Controls of Central and Peripheral Blood Pressure and Hemorrhagic/Hypovolemic Shock. J Clin Med. 2023 Jan 31;12(3):1108. doi: 10.3390/jcm12031108. PMID 36769755
- [Background] Chalkias A, Pais G, Gulati A. Effect of Centhaquine on the Coagulation Cascade in Normal State and Uncontrolled Hemorrhage: A Multiphase Study Combining Ex Vivo and In Vivo Experiments in Different Species. Int J Mol Sci. 2024 Mar 20;25(6):3494. doi: 10.3390/ijms25063494. PMID 38542464
- [Background] Khanna A, Vaidya K, Shah D, Ranjan AK, Gulati A. Centhaquine Increases Stroke Volume and Cardiac Output in Patients with Hypovolemic Shock. J Clin Med. 2024 Jun 27;13(13):3765. doi: 10.3390/jcm13133765. PMID 38999331
- [Background] Gulati A, Choudhuri R, Gupta A, Singh S, Ali SKN, Sidhu GK, Haque PD, Rahate P, Bothra AR, Singh GP, Maheshwari S, Jeswani D, Haveri S, Agarwal A, Agrawal NR. A Multicentric, Randomized, Controlled Phase III Study of Centhaquine (Lyfaquin(R)) as a Resuscitative Agent in Hypovolemic Shock Patients. Drugs. 2021 Jun;81(9):1079-1100. doi: 10.1007/s40265-021-01547-5. Epub 2021 Jun 1. PMID 34061314
- [Background] Gulati A, Jain D, Agrawal NR, Rahate P, Choudhuri R, Das S, Dhibar DP, Prabhu M, Haveri S, Agarwal R, Lavhale MS. Resuscitative Effect of Centhaquine (Lyfaquin(R)) in Hypovolemic Shock Patients: A Randomized, Multicentric, Controlled Trial. Adv Ther. 2021 Jun;38(6):3223-3265. doi: 10.1007/s12325-021-01760-4. Epub 2021 May 10. PMID 33970455
- [Background] Kontouli Z, Staikou C, Iacovidou N, Mamais I, Kouskouni E, Papalois A, Papapanagiotou P, Gulati A, Chalkias A, Xanthos T. Resuscitation with centhaquin and 6% hydroxyethyl starch 130/0.4 improves survival in a swine model of hemorrhagic shock: a randomized experimental study. Eur J Trauma Emerg Surg. 2019 Dec;45(6):1077-1085. doi: 10.1007/s00068-018-0980-1. Epub 2018 Jul 13. PMID 30006694
- [Background] Ranjan AK, Zhang Z, Briyal S, Gulati A. Centhaquine Restores Renal Blood Flow and Protects Tissue Damage After Hemorrhagic Shock and Renal Ischemia. Front Pharmacol. 2021 May 3;12:616253. doi: 10.3389/fphar.2021.616253. eCollection 2021. PMID 34012389
- [Background] Papalexopoulou K, Chalkias A, Pliatsika P, Papalois A, Papapanagiotou P, Papadopoulos G, Arnaoutoglou E, Petrou A, Gulati A, Xanthos T. Centhaquin Effects in a Swine Model of Ventricular Fibrillation: Centhaquin and Cardiac Arrest. Heart Lung Circ. 2017 Aug;26(8):856-863. doi: 10.1016/j.hlc.2016.11.008. Epub 2016 Dec 19. PMID 28385449
- [Background] O'Donnell JN, O'Donnell EP, Kumar EJ, Lavhale MS, Andurkar SV, Gulati A, Scheetz MH. Pharmacokinetics of centhaquin citrate in a dog model. J Pharm Pharmacol. 2016 Jun;68(6):803-9. doi: 10.1111/jphp.12554. Epub 2016 Apr 25. PMID 27109141
- [Background] O'Donnell JN, Gulati A, Lavhale MS, Sharma SS, Patel AJ, Rhodes NJ, Scheetz MH. Pharmacokinetics of centhaquin citrate in a rat model. J Pharm Pharmacol. 2016 Jan;68(1):56-62. doi: 10.1111/jphp.12498. Epub 2016 Jan 4. PMID 26725913
- [Background] Papapanagiotou P, Xanthos T, Gulati A, Chalkias A, Papalois A, Kontouli Z, Alegakis A, Iacovidou N. Centhaquin improves survival in a swine model of hemorrhagic shock. J Surg Res. 2016 Jan;200(1):227-35. doi: 10.1016/j.jss.2015.06.056. Epub 2015 Jun 29. PMID 26216751
- [Background] Gulati A, Zhang Z, Murphy A, Lavhale MS. Efficacy of centhaquin as a small volume resuscitative agent in severely hemorrhaged rats. Am J Emerg Med. 2013 Sep;31(9):1315-21. doi: 10.1016/j.ajem.2013.05.032. Epub 2013 Jul 19. PMID 23871440
- [Background] Lavhale MS, Havalad S, Gulati A. Resuscitative effect of centhaquin after hemorrhagic shock in rats. J Surg Res. 2013 Jan;179(1):115-24. doi: 10.1016/j.jss.2012.08.042. Epub 2012 Sep 2. PMID 22964270
- [Background] Gulati A, Lavhale MS, Garcia DJ, Havalad S. Centhaquin improves resuscitative effect of hypertonic saline in hemorrhaged rats. J Surg Res. 2012 Nov;178(1):415-23. doi: 10.1016/j.jss.2012.02.005. Epub 2012 Apr 2. PMID 22487389